CLINICAL TRIAL: NCT05083975
Title: Effect of Buzzy System (Vibrating Device) Compared to Topical Anaesthesia on Pain Reduction During Injection of Infiltration Anaesthesia in Children: A Randomized Clinical Trial.
Brief Title: Buzzy System Compared to Topical Anaesthesia During Infiltration Injection in Children.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Mahmoud Mohamed Mahmoud, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Buzzy System in Children.
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Local Anaesthesia
MeSH Terms: interventions — Anesthetics, Local; Carticaine; Epinephrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Both the patient and the investigator cannot be blinded due to the different techniques.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buzzy System (Experimental): Maxillary anesthetic infiltration injection using a conventional 2-ml syringe and a short needle after activating the buzzy device extra orally proximal to the site of injection for 30-60 seconds.
  Interventions: Device: Buzzy System; Drug: 1.8 ml of 4% articaine hydrochloride with epinephrine 1:100,000
- Control (Active Comparator): Maxillary anesthetic infiltration injection using a conventional 2-ml syringe and a short needle after application of 20% Benzocaine topical anesthestic gel.
  Interventions: Drug: Topical anesthetic; Drug: 1.8 ml of 4% articaine hydrochloride with epinephrine 1:100,000

INTERVENTIONS:
Device: Buzzy System — Vibrating Device
  Arms: Buzzy System
Drug: Topical anesthetic — 20% benzocaine gel (Opahl Topical Gel)
  Arms: Control
Drug: 1.8 ml of 4% articaine hydrochloride with epinephrine 1:100,000 — Local dental anesthetic agent

SUMMARY:
Aim of the study is to test the effect of Buzzy System (vibrating device) compared to topical anaesthesia on pain reduction during injection of infiltration anaesthesia in children.

ELIGIBILITY:
Inclusion Criteria:

1. Children classified as cooperative or potentially cooperative according to Wright's classification of child behaviour with rating 3 (positive) or 4 (definitely positive) according to Frankl behaviour rating scale.
2. Children aged 5-8 years old.
3. Patients who need maxillary buccal infiltration anesthesia.

Exclusion Criteria:

1. Children with any neurological or psychological disorders.
2. Children with known allergy to topical or local anesthetic agents.
3. Parental refusal for participation.
4. Children with previous history of local anesthesia injection.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2022-07-23 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
Pain Perception during local anaesthesia injection | Procedure (During and immediately after the administration of local anesthesia)
  Pain intensity directly after the injection recorded by Wong-Baker faces pain rating scale and Faces, Legs, Arms, Crying, Consolability (FLACC) scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Shilpapriya M, Jayanthi M, Reddy VN, Sakthivel R, Selvaraju G, Vijayakumar P. Effectiveness of new vibration delivery system on pain associated with injection of local anesthesia in children. J Indian Soc Pedod Prev Dent. 2015 Jul-Sep;33(3):173-6. doi: 10.4103/0970-4388.160343. PMID 26156269
- [Background] Hegde KM, R N, Srinivasan I, D R MK, Melwani A, Radhakrishna S. Effect of vibration during local anesthesia administration on pain, anxiety, and behavior of pediatric patients aged 6-11 years: A crossover split-mouth study. J Dent Anesth Pain Med. 2019 Jun;19(3):143-149. doi: 10.17245/jdapm.2019.19.3.143. Epub 2019 Jun 30. PMID 31338420
- [Background] Alanazi KJ, Pani S, AlGhanim N. Efficacy of external cold and a vibrating device in reducing discomfort of dental injections in children: A split mouth randomised crossover study. Eur Arch Paediatr Dent. 2019 Apr;20(2):79-84. doi: 10.1007/s40368-018-0399-8. Epub 2018 Dec 5. PMID 30519955
- [Background] Suohu T, Sharma S, Marwah N, Mishra P. A Comparative Evaluation of Pain Perception and Comfort of a Patient Using Conventional Syringe and Buzzy System. Int J Clin Pediatr Dent. 2020 Jan-Feb;13(1):27-30. doi: 10.5005/jp-journals-10005-1731. PMID 32581474
- [Background] AlHareky M, AlHumaid J, Bedi S, El Tantawi M, AlGahtani M, AlYousef Y. Effect of a Vibration System on Pain Reduction during Injection of Dental Anesthesia in Children: A Randomized Clinical Trial. Int J Dent. 2021 Jan 30;2021:8896408. doi: 10.1155/2021/8896408. eCollection 2021. PMID 33564311
- [Background] Faghihian R, Rastghalam N, Amrollahi N, Tarrahi MJ. Effect of vibration devices on pain associated with dental injections in children: A systematic review and meta-analysis. Aust Dent J. 2021 Mar;66(1):4-12. doi: 10.1111/adj.12811. Epub 2020 Dec 17. PMID 33258142
- [Background] Zielinski J, Morawska-Kochman M, Zatonski T. Pain assessment and management in children in the postoperative period: A review of the most commonly used postoperative pain assessment tools, new diagnostic methods and the latest guidelines for postoperative pain therapy in children. Adv Clin Exp Med. 2020 Mar;29(3):365-374. doi: 10.17219/acem/112600. PMID 32129952
- [Background] Hindocha N, Manhem F, Backryd E, Bagesund M. Ice versus lidocaine 5% gel for topical anaesthesia of oral mucosa - a randomized cross-over study. BMC Anesthesiol. 2019 Dec 16;19(1):227. doi: 10.1186/s12871-019-0902-8. PMID 31842771
- [Background] Al-Melh MA, Andersson L. Comparison of topical anesthetics (EMLA/Oraqix vs. benzocaine) on pain experienced during palatal needle injection. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 May;103(5):e16-20. doi: 10.1016/j.tripleo.2006.11.033. Epub 2007 Feb 27. PMID 17331753